CLINICAL TRIAL: NCT04920500
Title: A Randomized, Double-blind, Multiple-Dose, Two-Cycle, Parallel-Group, Bioequivalence Pretrial of Daunorubicin Cytarabine Liposome for Injection in Older, Naive AML Patients
Brief Title: Bioequivalence of Daunorubicin Cytarabine Liposomes in Naive AML Patients
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: CSPC Zhongnuo Pharmaceutical (Shijiazhuang) Co., Ltd. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: HC1702-BE-001
Record Dates: First submitted 2021-02-05; First posted 2021-06-09 (Actual); Last update posted 2021-06-09 (Actual); Status verified 2021-02

CONDITIONS: Acute Myeloid Leukemia
MeSH Terms: conditions — Leukemia, Myeloid, Acute | interventions — Injections

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Daunorubicin Cytarabine liposome for injection (Experimental): Induction 1: Daunorubicin Cytarabine liposome for injection [100 U/m²] i.v. (120 min±10min) d1,3,5 Induction 2: Daunorubicin Cytarabine liposome for injection [100 U/m²] i.v. (120 min±10min) d1,3 Consolidation therapy: Daunorubicin Cytarabine liposome for injection [65 U/m²] i.v. (>90 min) d1,3
  Interventions: Drug: Daunorubicin Cytarabine liposome for injection
- Vyxeos + Daunorubicin Cytarabine liposome for injection (Active Comparator): Induction 1: Vyxeos[100 U/m²] i.v. (120 min) d1; Daunorubicin Cytarabine liposome for injection [100 U/m²] i.v. (120 min±10min) d3,5 Induction 2: Daunorubicin Cytarabine liposome for injection [100 U/m²] i.v. (120 min±10min) d1,3 Consolidation therapy: Daunorubicin Cytarabine liposome for injection [65 U/m²] i.v. (>90 min) d1,3
  Interventions: Drug: Vyxeos、Daunorubicin Cytarabine liposome for injection

INTERVENTIONS:
Drug: Daunorubicin Cytarabine liposome for injection — Induction 1: [100 U/m²] i.v. d1,3,5 Induction 2: [100 U/m²] i.v. d1,3
  Arms: Daunorubicin Cytarabine liposome for injection
Drug: Vyxeos、Daunorubicin Cytarabine liposome for injection — Induction 1: [100 U/m²] i.v. Vyxeos（d1）,Daunorubicin Cytarabine liposome for injection（d3、d5） Induction 2: [100 U/m²] i.v. Daunorubicin Cytarabine liposome for injection（d1、d3 ）
  Other Names: Vyxeos
  Arms: Vyxeos + Daunorubicin Cytarabine liposome for injection

SUMMARY:
A Randomized, Double-blind, Multiple-Dose, Two-Cycle, Parallel-Group, Bioequivalence pretrial of Daunorubicin Cytarabine liposome for Injection in older, naive patients with Acute Myeloid Leukemia (AML).

DETAILED DESCRIPTION:
Bioequivalence Study of Daunorubicin Cytarabine liposome for injection, 100 units (CHINO Pharmaceutical Group Shijiazhuang Pharmaceutical Co Ltd), versus Vyxeos®, 100 units (Jazz Pharmaceuticals Public Limited Company), in patients with AML .

ELIGIBILITY:
Inclusion Criteria:

1. Patient volunteers to participate in this study and sign the informed consent form.
2. Aged 55-70 years, no gender limitation.
3. Patient has a diagnosis of untreated AML according to WHO criteria.
4. Eastern Cooperation Oncology Group (ECOG) performance status of 0~1.
5. Patient has a life expectancy of 3 months or longer.
6. Patients can be followed up as required by the study.
7. Patient must meet the following criteria as indicated on the clinical laboratory tests within 7 days prior to treatment :

   1. White Blood Cell Count≤ 50 x 10^9;
   2. Serum creatinine ≤ 1.5 x ULN
   3. Serum total bilirubin ≤ 1.5 x ULN; ≤3 x ULN in patients with liver infiltration
   4. Serum aspartate aminotransferase and alanine aminotransferase ≤ 2.5 x ULN;≤ 5 x ULN in patients with liver infiltration
   5. Coagulation function INR or PT ≤ 1.5 x ULN; APTT ≤ 1.5 x ULN
8. Left ventricular ejection fraction ≥ 50% as assessed by echocardiography or cardiac scan with multiple uptakes gated acquisition (MUGA).
9. Patients with mean value of triplicate Fridericia-corrected QT interval (QTcF) in the screening period, male < 450 ms, female < 470 ms.
10. Female or male patients of childbearing age agree to take effective contraception (such as intrauterine device [IUD], contraceptives or condoms) from the date of signing an informed consent to 180 days after the last dose and female patients must be non-lactating with a negative pregnancy test within 7 days.

Exclusion Criteria:

1. Patient has a diagnosis of acute promyelocytic leukemia (APL).
2. AML with central nervous system (CNS) involvement.
3. Patient has been previously diagnosed with another malignancy (except in the following cases: Patients with cured basal or squamous cell skin cancer, superficial bladder cancer, breast or cervical carcinoma in situ or focal prostate cancer with a Gleason score of 6).
4. Patient with prior exposures to daunorubicin or other anthracyclines, or cytarabine.
5. The interval between any treatment medication (conventional or investigational) for MDS and the first administration of this study is less than 2 weeks. However, the interval between the first medication of this study and hydroxyurea which used to inhibit the rapid proliferation of the tumor could be ≥ 24 hours. The study treatment should be held until the toxicity be reduced to Grade 1 or below.
6. Patients who have undergone major surgery or received radiotherapy within 4 weeks before the first study dose.
7. Patients who suffered from active cardiovascular diseases including but not limited to: poorly controlled hypertension (ie. systolic blood pressure ≥160 mmHg and/or diastolic blood pressure ≥ 90 mmHg ), myocardial infarction, unstable angina, uncontrolled arrhythmia, heart failure NYHA class III/IV within 6 months before the first study dose.
8. Patient has a history of severe bleeding, such as hemophilia A, hemophilia B, von Willebrand disease or spontaneous bleeding that requires blood transfusion or other medical intervention.
9. Patient has a history of stroke or intracranial hemorrhage within 6 months before the first study dose.
10. Patient has severe lung disease within 2 weeks before the first study dose.
11. Patient has an active uncontrolled infection (acute or chronic fungal, bacterial, viral or other infections).
12. Incapacity to give informed consent owe to any severe medical reasons, laboratory abnormalities or mental illness .
13. Patients who have severe allergic reactions or be intolerable to liposome preparation ingredients.
14. Patients with hepatolenticular degeneration or other abnormal copper metabolism.
15. Patients with positive hepatitis B surface antigen or hepatitis B core antibody with hepatitis B virus DNA > ULN by quantitative assay, positive hepatitis C antibody or positive HIV antibody.
16. Patients who have a special diet such as grapefruit within 48 hours before the first study dose.
17. Patients have received other clinical trial drugs within 28 days before screening.
18. Patients are not suitable for the study in the investigator's opinion.

Ages: 55 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 16 (Estimated)
Dates: Start 2020-09-04 (Actual); Primary Completion 2021-06-30 (Estimated); Study Completion 2021-06-30 (Estimated)

PRIMARY OUTCOMES:
Pharmacokinetics（PK） of Daunorubicin Cytarabine liposomes. | up to12 days
  Maximum concentration (Cmax) .
PK of Daunorubicin Cytarabine liposomes. | predose and up to 24 hours post-dose
  Area under the concentration curve at each cycle D1 (AUC0-24).

SECONDARY OUTCOMES:
Safety assessed by adverse events | up to 1 years
  An adverse event (AE) is defined as any untoward medical occurrence in a participant administered a study drug or has undergone study procedures and which does not necessarily have a causal relationship with this treatment. An AE can therefore be any unintended sign (including an abnormal laboratory finding), symptom or disease temporally associated with the use of a medicinal investigational) product, whether or not related to the medicinal (investigational) product.
Overall Response Rate (ORR) | up to 1 years
  The number and percentage of CR and CRi in each group were calculated

CONTACTS AND LOCATIONS:
Locations (1):
- Institute of Hematology and Hospital of Blood Disease, Chinese Academy of Medical Sciences, Tianjin, China